CLINICAL TRIAL: NCT06991894
Title: Real-world Outcomes of Aplastic Anemia Patients Treated With Eltrombopag: A Retrospective Medical Claims Database Study (Eltrombopag for Aplastic Anemia)
Brief Title: Real-world Outcomes of Aplastic Anemia Patients Treated With Eltrombopag: A Medical Claims Database Study
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CETB115EJP04
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Anemia, Aplastic
Keywords: Eltrombopag; Effectiveness; Safety; Treatment patterns
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Anatomical Therapeutic Chemical (ATG)-free Cohort: Japanese patients with AA from the MDV database who received treatment with ciclosporin A (CSA) alone, ETB alone, or a combination of CSA and ETB.
- ATG-Inclusive Cohort: Japanese patients with AA from the MDV database who received one of the following treatment combinations: CSA and ATG or CSA and ETB and ATG.

SUMMARY:
The main goal of this study was to investigate the effectiveness and safety of eltrombopag (ETB) when compared to other treatments in Japanese aplastic anemia (AA) patients using data from the Medical Data Vision (MDV) hospital-based database.

ELIGIBILITY:
Inclusion and exclusion criteria for the safety population:

Inclusion criteria:

* Patients with:

  * At least one confirmed diagnosis of AA registered during the baseline period, or
  * At least one confirmed diagnosis of idiopathic thrombocytopenic purpura (International Classification of Diseases, 10th Revision [ICD10] code: D69.3) registered before the index date and at least one confirmed diagnosis of AA during the follow-up period.
* Had at least 6 months of continuous enrolment prior to the index date.

Confirmed diagnosis was defined as having ≥1 inpatient or ≥2 outpatient claims with a relevant ICD-10 code and without any doubtful flag.

Continuous enrolment (being continuously followed in the database) was defined as having at least one claim every semester.

Exclusion Criteria:

* Not receiving ATG, CSA, ETB or romiplostim (ROM) during the selection period,
* Had a diagnosis of acute myeloid leukemia (AML), chronic myelomonocytic leukemia (CMML), myelofibrosis, other hematological malignancies, or cataract before the index date.

Inclusion and exclusion criteria for the effectiveness population:

Inclusion criteria:

* Had at least one confirmed diagnosis of AA registered before the index date,
* Had at least one procedure for any type of transfusion such as red blood cell transfusion, platelet transfusion, or granulocyte transfusion registered during the baseline period or within 4 weeks after the index date,
* Had at least 6 months of continuous enrolment prior to the index date,
* Had at least a 6-month follow-up period.

Exclusion criteria:

* Not receiving ATG, CSA, ETB or ROM during the selection period,
* Had at least one prescription of ATG, CSA, ETB or ROM before the index date,
* Had a diagnosis of AML, CMML or other hematological malignancies before the index date.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 2517 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Probability of Achieving Hematologic Response by AA Treatment Category | Month 6, Years 1, 2, and up to approximately 3 years
  The Kaplan-Meier analysis technique was used to estimate probability. Hematologic response was defined as the first occurrence of an 8-week period without any transfusion procedure. Treatment categories included:
  * CSA alone
  * CSA + ETB
  * ETB alone
  * ATG + CSA
  * ATG + CSA + ETB
Probability of Achieving Hematologic Response by ETB Dose Density | Month 6, Years 1, 2, and up to approximately 3 years
  The Kaplan-Meier analysis technique was used to estimate probability. Hematologic response was defined as the first occurrence of an 8-week period without any transfusion procedure. ETB dose density was defined as the dosage of ETB divided by the duration to maximum dose:
  * Optimal dose-density: 62.5 milligrams (mg) or more mg/8 weeks,
  * Suboptimal dose-density: 25.1-62.4 mg/8 weeks,
  * Minimum dose: 25 mg or less/8weeks.
Time to Achieve First Hematologic Response by AA Treatment Category | Up to approximately 3 years
  Time to hematologic response was defined as the number of days from the index date + 28 days to the first hematologic response. The index date was defined as the date of the first prescription of the following AA treatments: ATG, CSA, ETB or ROM. Event-free patients were censored at the earliest record of any of the following: death, end of the database registration, or end of the study. Treatment categories included:
  * CSA alone
  * CSA + ETB
  * ETB alone
  * ATG + CSA
  * ATG + CSA + ETB
Time to Achieve First Hematologic Response by ETB Dose Density | Up to approximately 3 years
  Time to hematologic response was defined as the number of days from the index date + 28 days to the first hematologic response. The index date was defined as the date of the first prescription of the following AA treatments: ATG, CSA, ETB or ROM. Event-free patients were censored at the earliest record of any of the following: death, end of the database registration, end of the study. ETB dose density was defined as the dosage of ETB divided by the duration to maximum dose:
  * Optimal dose-density: 62.5 mg or more mg/8 weeks,
  * Suboptimal dose-density: 25.1-62.4 mg/8 weeks,
  * Minimum dose: 25 mg or less/8weeks.
Percentage of Patients who Achieved Hematologic Response by Treatment Category | Months 3 and 6
  Hematologic response was defined as the first occurrence of an 8-week period without any transfusion procedure. Treatment categories included:
  * CSA alone
  * CSA + ETB
  * ETB alone
  * ATG + CSA
  * ATG + CSA + ETB
Cox Proportional Hazard Ratio for the Association Between Hematologic Response and Patient Characteristics | Up to approximately 3 years
  Patient characteristics included age, body mass index (BMI), treatment category (CSA+ETB vs CSA and ETB vs CSA), gender, comorbidity, medications received (antibiotics, anti-inflammatory drugs, anticonvulsants, antipsychotics), and bone marrow conditioning received before bone marrow transplant (BMT).

SECONDARY OUTCOMES:
Number of Patients per Demographic Category | Baseline
  Demographics included:
  * Age category
  * Gender
  * BMI
  * Most frequent comorbidities
  * Most frequent medications received
Hemoglobin Level | Baseline
Platelets Count | Baseline
Neutrophil Level | Baseline
Number of Blood Transfusions | Up to approximately 7 months
Total Units of Blood Transfusions | Up to approximately 7 months
Total Amount of Blood and Plasma Transfused | Up to approximately 7 months
Percentage of Patients With at Least One Transfusion of 400 Milliliters (mL) or More of red Blood Cells | Up to approximately 8 weeks
Percentage of Patients who Achieved Complete Response (CR) | Month 6
  CR was defined as hemoglobin >100 grams per liter (g/L) and neutrophils >1.0x10^9/L and platelets >100x10^9/L.
Percentage of Patients who Achieved Partial Response (PR) | Month 6
  PR was defined as no longer meeting severe AA criteria, transfusion independence, hemoglobin >8 grams per deciliter (gr/dL) and neutrophils >0.5x10^9/L and platelets >20x10^9/L.
Percentage of Patients who Achieved Overall Response | Month 6
  Overall response was defined as having CR or PR. CR was defined as hemoglobin >100 g/L and neutrophils >1.0x10^9/L and platelets >100x10^9/L. PR was defined as no longer meeting severe AA criteria, transfusion independence, hemoglobin >8 gr/dL and neutrophils >0.5x10^9/L and platelets >20x10^9/L.
Probability of Achieving an Effectiveness Event by Treatment Category | Month 6, Years 1, 2, and up to approximately 3 years
  The Kaplan-Meier analysis technique was used to estimate probability. Effectiveness events included death, treatment discontinuation, relapse, BMT, bleeding, bleeding requiring transfusion, bleeding requiring a treatment, and infection. Treatment categories included:
  * CSA alone
  * CSA + ETB
  * ETB alone
  * ATG + CSA
  * ATG + CSA + ETB
Probability of Achieving an Effectiveness Event by ETB Dose Density | Month 6, Years 1, 2, and up to approximately 3 years
  The Kaplan-Meier analysis technique was used to estimate probability. Effectiveness events included death, treatment discontinuation, relapse, BMT, bleeding, bleeding requiring transfusion, bleeding requiring a treatment, and infection. ETB dose density was defined as the dosage of ETB divided by the duration to maximum dose:
  * Optimal dose-density: 62.5 mg or more mg/8 weeks,
  * Suboptimal dose-density: 25.1-62.4 mg/8 weeks,
  * Minimum dose: 25 mg or less/8weeks.
Time to Achieve an Effectiveness Event by Treatment Category | Up to approximately 3 years
  Time to an effectiveness event was defined as the number of days from the index date + 28 days until the earliest record of an event of interest. The index date was defined as the date of the first prescription of the following AA treatments: ATG, CSA, ETB or ROM. Event-free patients were censored at the earliest record of any of the following: death, end of follow-up, or end of the study.
  Effectiveness events included death, treatment discontinuation, relapse, BMT, bleeding, bleeding requiring transfusion, bleeding requiring a treatment, and infection. Treatment categories included:
  * CSA alone
  * CSA + ETB
  * ETB alone
  * ATG + CSA
  * ATG + CSA + ETB
Time to Achieve an Effectiveness Event by ETB Dose Density | Up to approximately 3 years
  Time to an effectiveness event was defined as the number of days from the index date + 28 days until the earliest record of an event of interest. The index date was defined as the date of the first prescription of the following AA treatments: ATG, CSA, ETB or ROM. Event-free patients were censored at the earliest record of any of the following: death, end of follow-up, or end of the study.
  Effectiveness events included death, treatment discontinuation, relapse, BMT, bleeding, bleeding requiring transfusion, bleeding requiring a treatment, and infection. ETB dose density was defined as the dosage of ETB divided by the duration to maximum dose:
  * Optimal dose-density: 62.5 mg or more mg/8 weeks,
  * Suboptimal dose-density: 25.1-62.4 mg/8 weeks,
  * Minimum dose: 25 mg or less/8weeks.
Number of Patients who Received First Line Treatment by Type of Treatment Received | Up to approximately 3 years
Number of Patients who Received Second Line Treatment by Type of Treatment Received | Up to approximately 3 years
Number of Patients who Received Third Line Treatment by Type of Treatment Received | Up to approximately 3 years
Probability of Having a Safety Event by Treatment Category | Month 6, and Years 1, 2, and 5
  The Kaplan-Meier analysis technique was used to estimate probability. Safety events included diabetes, hepatotoxicity event, hypertension event, thromboembolic event, transformation to myelodysplastic syndrome (MDS), AML, CMML or other leukemia, and transformation to paroxysmal nocturnal hemoglobinuria (PNH).
  Treatment categories included:
  * CSA alone
  * CSA + ETB
  * ETB alone
  * ATG + CSA
  * ATG + CSA + ETB
Time to Having a Safety Event by Treatment Category | Up to approximately 9 years
  Time to each safety event was defined as the number of days from the index date until the earliest record of the event of interest. The index date was defined as the date of the first prescription of the following AA treatments: ATG, CSA, ETB or ROM. Event-free patients were censored at the earliest record of any of the following: death, end of follow-up, or end of the study.
  Safety events included diabetes, hepatotoxicity event, hypertension event, thromboembolic event, transformation to MDS, AML, CMML or other leukemia, and transformation to PNH.
  Treatment categories included:
  * CSA alone
  * CSA + ETB
  * ETB alone
  * ATG + CSA
  * ATG + CSA + ETB

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States